CLINICAL TRIAL: NCT04239534
Title: Continued Access Protocol For Convergence Of Epicardial And Endocardial RF Ablation For The Treatment Of Symptomatic Persistent AF CONVERGE CAP Study
Brief Title: CONVERGE CAP Study-For The Treatment Of Symptomatic Persistent or Long-standing Persistent AF
Acronym: CAP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Start-up and enrolling activities have been suspended and study closed
Sponsor: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP2019-1
Record Dates: First submitted 2020-01-13; First posted 2020-01-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2021-08

CONDITIONS: Atrial Fibrillation
Keywords: Hybrid Procedure
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Continued Access Protocol (CAP), prospective, multi-center, single arm study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Arm (Other): In this Single Arm Study, Epicardial linear lesions will be created endoscopically using the EPi-Sense-AF Guided Coagulation System with VisiTrax throughout the posterior left atrium and along the pericardial reflections from a trans-diaphragmatic or sub-xyphoid access. Followed by the sue of an endocardial ablation catheter that will be used to ablate endocardially to connect lesions at the reflections, complete the isolation of the pulmonary veins and create a cavotricuspid lesion to prevent typical atrial flutter.
  Interventions: Device: Convergence Of Epicardial And Endocardial RF Ablation

INTERVENTIONS:
Device: Convergence Of Epicardial And Endocardial RF Ablation — The epicardial lesion pattern will be created using the EPi-Sense®-AF Guided Coagulation System with VisiTrax®. Epicardial linear lesions will be created endoscopically using the EPi-Sense-AF Guided Coagulation System with VisiTrax throughout the posterior left atrium and along the pericardial reflections from a trans-diaphragmatic or sub-xyphoid access without any chest incisions. An endocardial ablation catheter will be used to ablate endocardially to connect lesions at the reflections, complete the isolation of the pulmonary veins and create a cavotricuspid lesion to prevent typical atrial flutter. Once the study lesion pattern has been created by coagulating cardiac tissue using the EPi- Sense-AF Guided Coagulation System and the endocardial ablation catheter, the pulmonary veins must be evaluated for entrance and/or exit block to confirm isolation.

SUMMARY:
The objective of this clinical study is to collect additional data on the safety and effectiveness of the EPi- Sense®-AF Guided Coagulation System with VisiTrax® to treat symptomatic persistent or long-standing persistent Atrial Fibrillation (AF) patients who are refractory or intolerant to at least one Class I and/or III AAD.

DETAILED DESCRIPTION:
This is a prospective CAP, multi-center, single arm study. The study will enroll one hundred and seventy subjects (170) to ensure that 153 subjects are treated with the EPi-Sense®-AF device, after accounting for post-enrollment subject ineligibility. Patients will be enrolled from up to twenty-seven (27) sites that enrolled patients in the CONVERGE study. For consistency, the same endpoints defined in the CONVERGE study will be used in the CAP.

The population for this study will be subjects with Persistent or Long-standing Persistent atrial fibrillation defined in accordance with the Heart Rhythm Society (HRS) 2017 AF expert consensus statement.

* Persistent: Continuous AF which is sustained beyond seven days.
* Long-standing Persistent: Continuous AF of greater than 12 months' duration. Subject informed consent might be obtained in two phases to allow for additional testing, beyond the site's standard of care (SOC) needed to complete the subject's eligibility to participate in this trial. If additional tests are needed to determine study eligibility, the subjects will sign a Screening ICF. Following a full evaluation, if it is determined that the subject is eligible to participate in the CONVERGE CAP study, the subject will sign an Enrollment ICF. Sites will continue to monitor subjects implanted with a loop recorder who did not qualify to be enrolled in the study. If the ILR indicates a change in the subject's AF status from paroxysmal to persistent AF and the subject continues to meet study eligibility criteria, the subject could sign an Enrollment consent to participate in the study.

Subjects will be provided the IRB/EC approved ICFs (Screening and Enrollment) and will have the opportunity to read, understand, and have their questions answered prior to signing the ICFs. If the subject agrees to participate in the study and signs consent, the ICF process will be completed. The subject must sign and date the Screening ICF prior to any additional assessments needed to determine study eligibility and sign and date the Enrollment ICF prior to study-specific procedures being performed. The person reviewing the ICF with the subject will also sign and date the ICFs. The subject will be given copies of the signed ICFs to keep. The Screening ICF will be required only if non-study evaluations are needed to determine the subject's eligibility to participate in the study.

Upon entering subject enrollment information into Clindex, each subject will be assigned a unique identification (ID) number sequentially in ascending order. All subjects who sign the ICFs will be documented in a Screening and Enrollment Log. For subjects who sign the Screening ICF but are ineligible to participate, minimum baseline characteristics: age, gender, race, screening date and screen failure reason (s) will be captured in Clindex.

Subjects are considered to be enrolled in the study when they have signed the Enrollment ICF. Subjects are considered to be treated when any of the study devices are introduced into the body.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and < 80 years at time of enrollment consent.
2. Left atrium ≤ 6.0 cm (Trans Thoracic Echo - TTE - parasternal 4 chamber view) or equivalent test.
3. Refractory or intolerant to at least one AAD (class I and/or III).
4. Subject has history of persistent or long-standing persistent atrial fibrillation as defined by the 2017 HRS/EHRA/ECAS Guidelines.
5. Provided written informed consent.

Exclusion Criteria:

1. Patients requiring concomitant surgery such as valvular repair or replacement, coronary artery bypass graft (CABG) surgery and atrial septal defect closure.
2. Left ventricular ejection fraction < 40%.
3. Pregnant or planning to become pregnant during study.
4. Co-morbid medical conditions that limit one-year life expectancy.
5. Previous cardiac surgery.
6. History of pericarditis.
7. Previous cerebrovascular accident (CVA), excluding fully resolved TIA.
8. Patients who have active infection or sepsis.
9. Patients with esophageal ulcers strictures and varices.
10. Patients with renal dysfunction who are not on dialysis (defined as GFR ≤ 40).
11. Patients who are contraindicated for anticoagulants such as heparin and coumadin.
12. Patients who are being treated for ventricular arrhythmias.
13. Patients who have had a previous left atrial catheter ablation for AF (does not include ablation for AFL or other supraventricular arrhythmias).
14. Patients with existing ICDs.
15. Current participation in another clinical investigation of a medical device or a drug, or recent participation in such a study within 30 days prior to study enrollment.
16. Not competent to legally represent him or herself (e.g., requires a guardian or caretaker as a legal representative).
17. Patient has presence of thrombus in the left atrium determined by intraoperative TEE.
18. Patient exhibits pulmonary vein stenosis in one or more of the pulmonary veins >50 % stenosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint- Freedom from Atrial Fibrillation, Atrial Tachycardia and Atrial Flutter | From Three month blanking period until 12-months post procedure follow-up visit.
  The primary effectiveness endpoint is freedom from AF/AT/AFL absent class I and III AADs except for a previously failed or intolerant class I or III AAD with no increase in dosage following the 3-months blanking period through the 12-months post procedure follow-up visit.
  The primary effectiveness endpoint will be evaluated from the 24-hours Holter.
Primary Safety Endpoint- Evaluation of major adverse events (MAEs) from the procedure to 30-days post procedure. | From procedure to 30-days post procedure
  The primary safety endpoint for the study is the incidence of major adverse events (MAEs) for subjects undergoing the convergent procedure from the procedure to 30-days post procedure. The following MAEs occurring within 30 days of the procedure will contribute toward the primary safety endpoint: cardiac tamponade, severe pulmonary vein (PV) stenosis, excessive bleeding, myocardial infarction, Stroke, transient ischemic attacks (TIA), atrioesophageal fistula (AEF), phrenic nerve injury, and death.

SECONDARY OUTCOMES:
Effectiveness-Freedom for Atrial Fibrillation, Atrial Tachycardia, Atrial Flutter and reduction of Atrial Fibrillation burden | From 3-month blanking to 12-, 24- and 36- months post procedure evaluation
  1. Freedom from AF/AT/AFL > 30 seconds in duration in the absence class I and III AADs except for a previously failed or intolerant class I or III AAD with no increase in dosage following the 3-months blanking period through the 24- and 36- months post procedure follow-up visits.
  2. Freedom from AF/AT/AFL > 1 hour in duration in the absence of class I and III AADs except for a previously failed or intolerant class I or III AAD with no increase in dosage following the 3-months blanking period through the 24 and 36- months post procedure follow-up visits.
Effectiveness- Atrial Fibrillation burden reduction | From 3-month blanking to 12-, 24- and 36- months post procedure evaluation
  1. Burden reduction of ≥75% and ≥90% from baseline AF burden and off all Class I and III AADs at 12, 24, and 36-months post procedure.
  2. Burden reduction of ≥75% and ≥90% from baseline AF burden regardless of Class I and III AAD status at 12, 24, and 36-months post procedure.
Safety-Incidence of serious adverse events | Through 12-months post procedure visit
  Incidence of serious adverse events (SAEs) in the study through the 12-months post procedure visit.

CONTACTS AND LOCATIONS:
Overall Officials: David De Lurgio, M.D., Principal Investigator — Emory University
Locations (10):
- United States (8):
  - Grandview Medical Center, Birmingham, Alabama
  - Heart Center Research LLC, Huntsville, Alabama
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - St. Vincent's HealthCare, Jacksonville, Florida
  - Palm Beach Gardens Medical Center, Palm Beach Gardens, Florida
  - Emory University - St. Joseph's Hospital, Atlanta, Georgia
  - Cardiology Associates Research, LLC, Tupelo, Mississippi
  - Virginia Cardiovascular Specialists, Richmond, Virginia
- United Kingdom (2):
  - St. Bartholomew's Hospital, London
  - Guy's and St. Thomas Hospital, London

IPD SHARING:
Plan to Share IPD: No